CLINICAL TRIAL: NCT01443182
Title: Treatment of PTSD in Adult Survivors of Early Chronic Interpersonal Trauma
Brief Title: Treatment of Posttraumatic Stress Disorder (PTSD) in Adult Survivors of Early Chronic Interpersonal Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL31098.097.10
Record Dates: First submitted 2011-09-27; First posted 2011-09-29 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAIR + MPE (Experimental): A two-phased treatment with Skills Training in Affective and Interpersonal Regulation (STAIR) in Phase 1 en modified prolonged exposure (MPE) in Phase 2
  Interventions: Behavioral: STAIR; Behavioral: MPE
- STAIR + EMDR (Active Comparator): a two-phase treatment Phase 1: Skills Training in Affective and Interpersonal Regulation (STAIR) Phase 2: Eye Movement Desensitization and Reprocessing (EMDR)
  Interventions: Behavioral: STAIR; Behavioral: EMDR

INTERVENTIONS:
Behavioral: STAIR — Skills Training in Affective and Interpersonal Regulation
Behavioral: MPE — Modified prolonged exposure (MPE)
  Arms: STAIR + MPE
Behavioral: EMDR — Eye movement desensitization and reprocessing
  Arms: STAIR + EMDR

SUMMARY:
Eye movement desensitization and reprocessing (EMDR) and trauma-focused cognitive-behavioural therapy (TF-CBT) have both been found to be effective in treating post-traumatic stress disorder (PTSD) following single-event traumas and to be more effective than pure anxiety management or stabilization treatments. However, much less is known about the efficacy of the different treatment approaches in survivors of repeated or chronic interpersonal trauma. Recent evidence suggests that a combination of stabilization treatment + TF-CBT is efficacious in this population. Although EMDR is also often used in survivors of chronic interpersonal trauma, evidence on its efficacy are still poor. The aim of the current study is to compare the efficacy of (1) stabilization + TF-CBT and (2) stabilization + EMDR using a randomized controlled trial in a routine clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* meeting DSM-IV criteria for PTSD
* having experienced repeated or chronic interpersonal trauma (e.g., sexual or physical abuse)
* at least 18 years of age
* having sufficient fluency in Dutch to complete treatment and research protocol
* participants using prescribed anti-depressant medication are required to be on a stable dose for at least 2 weeks before the beginning of treatment and remain on this dose throughout the treatment.

Exclusion Criteria:

* psychiatric problems that may interfere with the study participation or that require more intensive care than can be offered in the present study, including dementia, psychotic symptoms, depression with suicidal ideation, full-blown borderline personality disorder, substance dependence
* current use of tranquilizers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | Pre- (baseline) and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))
Posttraumatic Diagnostic Scale (PDS) | Pre- (baseline) and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up). Before each treatment session

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Pre- (baseline), after the first 8 treatment sessions and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))
Beck Anxiety Inventory (BAI) | Pre- (baseline), after the first 8 treatment sessions and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))
Dissociative Experiences Scale (DES) | Pre- (baseline), after the first 8 treatment sessions and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))
Difficulties in Emotion Regulation Scale (DERS) | Pre- (baseline), after the first 8 treatment sessions and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))
Inventory of Interpersonal Problems (IIP) | Pre- (baseline), after the first 8 treatment sessions and post-assessment (after treatment termination) and 3 month follow up (3 month after post assessment and 12 month follow up))

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ehring, PhD, Study Chair — University of Amsterdam; Katharina Meyerbröker, Study Chair — University of Amsterdam
Locations (1):
- PsyQ, Zaandam, Netherlands

REFERENCES:
- [Derived] Wigard I, Meyerbroker K, Ehring T, Topper M, Arntz A, Emmelkamp P. Skills training followed by either EMDR or narrative therapy for posttraumatic stress disorder in adult survivors of childhood abuse: a randomized controlled trial. Eur J Psychotraumatol. 2024;15(1):2332104. doi: 10.1080/20008066.2024.2332104. Epub 2024 Apr 17. PMID 38629403